CLINICAL TRIAL: NCT03515096
Title: Eltrombopag vs. Recombinant Human Thrombopoietin to Increase Platelet Level After Hematopoietic Stem Cell Transplantation: a Non-inferiority, Open-label, Randomized-controlled Study
Brief Title: Eltrombopag vs. rhTPO to Increase Platelet Level After HSCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201803070044
Record Dates: First submitted 2018-04-22; First posted 2018-05-03 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-06

CONDITIONS: Eltrombopag; Hematopoietic Stem Cell Transplantation; Thrombocytopenia
Keywords: rhTPO; HSCT; Thrombopoietin
MeSH Terms: conditions — Thrombocytopenia; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eltrombopag (Experimental): Thrombopoietin- receptor (TPO-R) agonist
  Interventions: Drug: Eltrombopag
- rhTPO (Placebo Comparator): Recombinant human thrombopoietin (rhTPO)
  Interventions: Drug: rhTPO

INTERVENTIONS:
Drug: Eltrombopag — Eltrombopag 50 mg; po; from day 1 to platelet is completely effective recovered after HSCT.
  Other Names: Promacta; Revolade
  Arms: Eltrombopag
Drug: rhTPO — rhTPO 15000 u; subcutaneously injection; from day 1 to platelet is completely effective recovered after HSCT.
  Other Names: no other name
  Arms: rhTPO

SUMMARY:
The primary objective is to compare the efficacy of eltrombopag vs rhTPO in complete response in patients after HSCT in China. This is a post-marketing, interventional, single-center, double-arm, prospective, open-label, non-inferior, randomized controlled study in adult patients with hematopoietic stem cell transplantation in China. Patients will be recruited consecutively from the study sites during the enrollment period. The enrolled patients will be given eltrombopag or rhTPO under the conditions of informed consent and frequent monitoring according to the clinical guideline.

DETAILED DESCRIPTION:
Hematopoietic stem cell transplantation (HSCT) is an important method to treat malignant tumor of blood system, and promoting platelets after HSCT is one of the important factors to determine the success of transplantation.

Recently, the main effective method to treat thrombocytopenia after transplantation is to preventively transfuse platelets. However, this method can cause platelet transfusion related graft-versus-host disease(GVHD), increase the risk of reaction and infection associated with blood transfusion, easily produce platelet related and specific antibodies (HPA), which seriously affect the curative effect of platelet infusion and even render platelet transfusion invalid. Besides, study has shown that the effective rate of platelet transfusion is 30%-70%, and the application of platelets in clinic is limited because of the shortage of blood supply at present.

Recombinant human thrombopoietin (rhTPO) is a glycoprotein molecule modified by full-length glycosylation and is of a similar pharmacological effect with endogenous thrombopoietin (TPO). TPO is a specific cytokine of megakaryocyte, which can promote the proliferation and maturation of macronuclear progenitor cells by binding to the receptor c-mpl. In addition, the chinese State Food and Drug Administration (SFDA) approved rhTPO for the treatment of thrombocytopenia after tumor chemotherapy in 2006. The study shows that rhTPO can increase the mean value of platelet count in the low period of platelet, shorten the time of low platelet, and improve the peripheral blood platelet aggregation rate in the bone marrow depression period.

Eltrombopag is the first oral non-peptide receptor (TPO-R) agonist, which can induce the proliferation and maturation of macronuclear progenitor cells via the Janus kinase (JAK) /signal transducer and activator of transcription (STAT) pathway. In 2008, the U.S. FDA approved the use of eltrombopag for the treatment of chronic idiopathic thrombocytopenia, and it has been widely used in tumor patients with thrombocytopenia after chemotherapy. Tanaka et al. have proved that eltrombopag can improve the average elevation of the platelet count in the bone marrow depression period in patients with stem cell transplantation. Besides, within the 9 patients receiving transplantation, the complete response of patients with primary and secondary thrombocytopenia were 60% and 71% respectively.

In China, studies showed that rhTPO could promote the recovery of platelet count, effectively reduce the infusion of platelet, decrease the risk of transplanting hemorrhage in acute leukemia patients after allo-HSCT. However, it is not clear that the effect of eltrombopag on improving platelet count after the treatment of HSCT. In addition, the comparison of efficacy and safety of eltrombopag vs rhTPO on platelet recovery after HSCT in clinical trial is not investigated. Therefore, it is of great significance to explore the efficacy and safety of eltrombopag and rhTPO in improving the recovery of platelet count after HSCT, which will provide a better method to recover platelet after HSCT.

The purpose of this study is to compare the efficacy of Eltrombopag vs rhTPO in complete response in patients after HSCT in China. To be more precise, Eltrombopag is taken 50 mg po daily from day 1 until platelet is completely effectively recovered after HSCT, while rhTPO is given by subcutaneous injection 15000 u daily from day 1 until platelet is completely effectively recovered after HSCT.

The primary endpoint was cumulative numbers of platelet engraftment (platelet recovery to ≥20 X 109/L for seven consecutive days without transfusion) on day 60 after transplantation

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18;
* Patients who have undergone hematopoietic stem cell transplantation (HSCT);
* Patients who don't take any drug including Eltrombopag and rhTPO before hematopoietic stem cell transplantation (HSCT);
* Patients receiving either an autologous (Auto) or allogeneic (Allo) stem cell transplantation from a sibling,related donor, or matched unrelated donor are included;
* Agree to sign informed consent

Exclusion Criteria:

* Patients with thrombocytopenia causes by other reasons, such as drugs, cytomegalovirus or infection;
* Patients who had greater risk of thromboembolic disease within six months;
* Patients with a history of heart disease;
* Patients with severe organ dysfunction;
* Patients with other malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2021-08-02 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
The cumulative numbers of platelet engraftment (platelet recovery to ≥20 X 109/L for seven consecutive days without transfusion) on day 60 after transplantation | From the start of study treatment (Day 1) to day 60

SECONDARY OUTCOMES:
Number of Participants (Responders) Achieving a Platelet Count >=30×10^9/L On Day 21 After HSCT | From the start of study treatment (Day 1) to days 21
  On days 21 after HSCT, the number of participants (responders) with platelet count >=30x10^9/L and no platelet infusion for 7 days were compared between treatments
Number of Participants (Responders) Achieving a Platelet Count >=100×10^9/L On Day 21 After HSCT | From the start of study treatment (Day 1) to days 21
  On days 21 after HSCT, the number of participants (responders) with platelet count >=100x10^9/L and no platelet infusion for 7 days were compared between treatments
Number of Participants With Bleeding events as Assessed Using the predefined bleeding scoring system. | From the start of study treatment (Day 1) to days 90
  The predefined bleeding scoring system is a measure of bleeding severity with the following score: score 0 = no bleeding, score 1= occult blood in body secretions (detected by heme-positive dipstick), mild petechiae, or minimal vaginal spotting, score 2= minor bleeding that does not require red blood cells (RBC) transfusions over routine transfusion needs (epistaxis, vaginal bleeding, mild hematemesis, melena, and mild hematuria) 3 = hemorrhage causing rapid decrease in hematocrit level, necessitating one or more units of RBCs per day beyond routine transfusion needs, and score 4 = Life-threatening hemorrhage, defined as either massive bleeding causing severe hemodynamic compromise or bleeding into vital organ (e.g., intracranial hemorrhage, pericardial, or diffuse alveolar hemorrhage).
Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE) | From the start of study treatment (Day 1) to days 90
  An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product.A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, is a congenital anomaly/birth defect or is associated with protocol specified liver injury and impaired liver function or is any protocol specific AEs.

CONTACTS AND LOCATIONS:
Overall Officials: XIN DU, MD, Principal Investigator — Second People's Hospital of Shenzhen
Locations (1):
- Shenzhen Second People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wen B, Zhang X, Chen S, Fan J, Yang S, Cai Y, Wang P, Zhang Q, Gu Q, Du X. Oral eltrombopag versus subcutaneous recombinant human thrombopoietin for promoting platelet engraftment after allogeneic stem cell transplantation: A prospective, non-inferiority, randomized controlled trial. Hematol Oncol. 2022 Oct;40(4):777-786. doi: 10.1002/hon.3017. Epub 2022 May 18. PMID 35554955